CLINICAL TRIAL: NCT00797511
Title: Immunogenicity and Safety of ADACEL POLIO (TdcP-IPV Vaccine) Administered at 6 to 8 Years of Age as a Fifth Dose in Healthy Children in Taiwan
Brief Title: Immunogenicity and Safety of Adacel Polio Vaccine
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: TD525
Record Dates: First submitted 2008-11-24; First posted 2008-11-25 (Estimated); Results first posted 2012-11-26 (Estimated); Last update posted 2012-11-26 (Estimated); Status verified 2012-10

CONDITIONS: Diphtheria; Tetanus; Pertussis; Poliomyelitis
Keywords: Diphtheria; Tetanus; Pertussis; Poliomyelitis
MeSH Terms: conditions — Diphtheria; Tetanus; Whooping Cough; Poliomyelitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Study Group (Experimental): Participants will receive one dose of Tetanus, diphtheria (reduced antigen content), pertussis (acellular components) vaccine (TdcP-IPV, ADACEL Polio) on Day 0
  Interventions: Biological: TdcP-IPV vaccine

INTERVENTIONS:
Biological: TdcP-IPV vaccine — 0.5 mL, Intramuscular
  Other Names: ADACEL POLIO

SUMMARY:
The present study is designed to meet the requirements of the Taiwanese Health Authorities for registration of ADACEL POLIO in Taiwan.

Subjects will receive one dose of the study vaccine at 6 to 8 years of age. Blood samples will be taken for antibody titration. The expected total duration of follow-up for each subject will be 28 days.

ELIGIBILITY:
Inclusion Criteria:

* Aged 6 to 8 years on the day of inclusion
* Informed consent form signed by the parent(s) or another legally acceptable representative
* Subject and parent/guardian able to attend all scheduled visits and comply with all trial procedures
* Written documentation of complete primary series and fourth dose of diphtheria, tetanus, pertussis (DTP) and Polio vaccines
* Parent(s)/legal representative present or fully completed pre-inclusion medical questionnaire.

Exclusion Criteria:

* Participation in another clinical trial investigating a vaccine, drug, medical device, or a medical procedure in the 4 weeks preceding the trial vaccination
* Planned participation in another clinical trial during the present trial period
* Known or suspected congenital or acquired immunodeficiency, immunosuppressive therapy such as anti-cancer chemotherapy or radiation therapy within the preceding 6 months, or long-term systemic corticosteroids therapy
* Known systemic hypersensitivity to any of the vaccine components (or residues carried over from manufacture, such as formaldehyde, glutaraldehyde, streptomycin, neomycin and polymyxin B ) or history of a life-threatening reaction to the trial vaccine or to a vaccine containing any of the same substances with specific focus on subjects who had, after previous administration of DTP vaccine, one of the pre-listed adverse events.
* Chronic illness, at a stage that could interfere with trial conduct or completion, in the opinion of the investigator
* Progressive neurologic disorder, including infantile spasms, uncontrolled epilepsy, progressive encephalopathy
* Receipt of blood or blood-derived products in the past 3 months, that might interfere with the assessment of immune response
* Receipt of any vaccine in the 4 weeks preceding the trial vaccination
* Planned receipt of any vaccine in the 4 weeks following the trial vaccination
* Known Human Immunodeficiency Virus (HIV), Hepatitis B surface (HBs) antigen, or Hepatitis C seropositivity
* History of diphtheria and/or tetanus and/or pertussis and/or poliomyelitis infection (confirmed either clinically, serologically or microbiologically)
* Previous fifth vaccination against diphtheria and/or tetanus and/or pertussis and/or poliomyelitis diseases with either the trial vaccine or another vaccine
* Thrombocytopenia, bleeding disorder or anticoagulants in the 3 weeks preceding inclusion contraindicating intramuscular (IM) vaccination
* Subject at high risk for diphtheria and/or tetanus and/or pertussis and/or poliomyelitis infection during the trial
* Received oral or injected antibiotic therapy within the 72 hours prior to any blood draw
* Febrile illness (temperature ≥ 37.5°C) or moderate or severe acute illness/infection on the day of vaccination, according to investigator judgment

Ages: 6 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 132 (Actual)
Dates: Start 2008-11; Primary Completion 2009-04 (Actual); Study Completion 2009-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Sanofi Pasteur Inc.
Locations (1):
- Taipei, Taipei, Taiwan

REFERENCES:
- See also: Related Info — http://www.sanofipasteur.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled from 24 November 2008 to 11 March 2009 at 1 medical center in Taiwan.
Pre-assignment Details: A total of 132 participants who met the inclusion and none of the exclusion criteria were enrolled, vaccinated, and evaluated.
Groups:
- ADACEL POLIO Vaccine Study Group: Participants received one dose of TdcP-IPV vaccine (ADACEL Polio) on Day 0.
Period: Overall Study
Arm/Group | ADACEL POLIO Vaccine Study Group
Started | 132
Completed | 131
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Groups:
- ADACEL POLIO Vaccine Study Group: Participants received one dose of Tetanus, diphtheria (reduced antigen content), pertussis (acellular components) vaccine (TdcP-IPV, ADACEL Polio) on Day 0
Arm/Group | ADACEL POLIO Vaccine Study Group
Number analyzed (Participants) | 132
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 132
  Between 18 and 65 years | 0
  >=65 years | 0
Age Continuous [Mean (Standard Deviation); unit: Years] | 6.89 (0.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 64
  Male | 68
Region of Enrollment [Number; unit: participants]
  Taiwan | 132

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Seroprotection to Vaccine Antigens Following Vaccination With ADACEL Polio (TdcP-IPV) Vaccine.
Description: Diphtheria concentrations determined by diphtheria toxin neutralization assay (Dip SN); Tetanus concentrations determined by enzyme-linked immunosorbent assay (ELISA).
  Seroprotection titer levels were defined as: Anti-diphtheria antibody titers ≥0.1 international unit (IU) per milliliter (mL); Anti-tetanus antibody titers ≥0.01 IU/mL and ≥0.1 IU/mL; Anti-Polio (≥ 8 1/dilution).
Time Frame: Day 28 post-vaccination
Population: Anti-tetanus and anti-diphtheria concentrations were assessed in the per-protocol population.
Measure: Number; unit: Participants
Arm/Group | ADACEL POLIO Vaccine Study Group
Number analyzed (Participants) | 131
Participants
  Anti-Diphtheria (Post-vaccination) | 131
  Anti-Tetanus (Post-vaccination) | 131
  Anti-Polio 1 (Post-vaccination) | 131
  Anti-Polio 2 (Post-vaccination) | 131
  Anti-Polio 3 (Post-vaccination) | 131

2. Primary Outcome: Number of Participants With Booster Response to Vaccine Pertussis Antigens Following Vaccination With ADACEL Polio (TdcP-IPV) Vaccine.
Description: The anti-Pertussis concentration were determined by ELISA. The criteria for demonstrating booster response are: (i) Pre-vaccination antibody concentrations less than the lower limit of quantitation (LLOQ) for each anti-pertussis antibody (PT, FHA, FIM, and PRN) but a post-vaccination levels ≥ 4 x LLOQ; or (ii) Pre-vaccination antibody concentrations ≥ LLOQ but < 4 x LLOQ with a 4-fold rise rate; or (iii) Pre-vaccination antibody concentrations ≥ 4 x LLOQ but with a 2-fold rise rate.
Time Frame: Day 28 post-vaccination
Population: Anti-Pertussis concentrations were assessed in the per-protocol population.
Measure: Number; unit: Participants
Groups:
- ADACEL POLIO Vaccine Study Group: Participants received a dose of Tdap or Tdap-vIPV vaccine on Day 0
Arm/Group | ADACEL POLIO Vaccine Study Group
Number analyzed (Participants) | 131
Participants
  Anti-Pertussis (N = 114) | 88
  Anti-Filamentous Hemagglutinin (N = 130) | 126
  Anti-Fimbriae types 2 and 3 (N = 130) | 116
  Anti-Pertactin (N = 131) | 130

3. Primary Outcome: Geometric Mean Titers (GMTs) of Antibodies to ADACEL Polio Vaccine Antigens Following Vaccination
Description: Diphtheria antibody concentrations determined by diphtheria toxin neutralization assay; Tetanus antibody concentrations determined by enzyme-linked immunosorbent assay (ELISA).
Time Frame: Day 28 post-vaccination
Population: Geometric mean titers were assessed in the per-protocol population.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | ADACEL POLIO Vaccine Study Group
Number analyzed (Participants) | 131
Titers
  Anti-Diphtheria (Post-vaccination) | 3.81 [3.25 to 4.46]
  Anti-Tetanus (Post-vaccination) | 17.2 [14.8 to 20.0]
  Anti-Polio 1 (Post-vaccination) | 9627 [7960 to 11642]
  Anti-Polio 2 (Post-vaccination) | 7083 [6057 to 8282]
  Anti-Polio 3 (Post-vaccination) | 9860 [8244 to 11793]

4. Primary Outcome: Geometric Mean Titers of Antibodies to Pertussis Antigens Following Vaccination With ADACEL Polio
Description: Pre- and post-vaccination GMTs for the Pertussis toxoid (PT), Pertussis filamentous hemagglutinin (FHA), Pertussis pertactin (PRN), and Pertussis Fimbriae types 2 and 3 (FIM), all determined by enzyme-linked immunosorbent assay (ELISA).
Time Frame: Day 0 (pre-vaccination) and Day 28 post-vaccination
Population: Geometric mean titers to the vaccine Pertussis antigens were assessed in the per-protocol population.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | ADACEL POLIO Vaccine Study Group
Number analyzed (Participants) | 131
Titers
  Anti-Pertussis Toxoid (Pre-vaccination) | 4.53 [3.81 to 5.39]
  Anti-Pertussis Toxoid (Post-vaccination) | 42.7 [36.1 to 50.3]
  Anti-Filamentous hemagglutinin (Pre-vaccination) | 19.7 [16.4 to 23.7]
  Anti-Filamentous hemagglutinin (Post-vaccination) | 164 [145 to 185]
  Anti-Fimbriae types 2 and 3 (Pre-vaccination) | 17.5 [12.8 to 24.0]
  Anti-Fimbriae types 2 and 3 (Post-vaccination) | 423 [291 to 614]
  Anti-Pertactin (Pre-vaccination) | 11.9 [9.92 to 14.3]
  Anti-Pertactin (Post-vaccination) | 314 [263 to 376]

5. Secondary Outcome: Number of Participants Reporting at Least 1 Solicited Injection Site or Systemic Reaction Post-vaccination With ADACEL Polio Vaccine
Description: Solicited Injection Site Reactions: Pain, Erythema/redness, Swelling, and Extensive swelling of vaccinated limb. Solicited Systemic Reactions: Fever (temperature ≥ 37.5ºC), Headache, Malaise, and Myalgia.
Time Frame: Day 0 up to Day 7 post-vaccination
Population: Safety analysis was on all enrolled and vaccinated participants with available reaction data, intent-to-treat population.
Measure: Number; unit: Participants
Arm/Group | ADACEL POLIO Vaccine Study Group
Number analyzed (Participants) | 132
Participants
  Any Solicited Injection Site Reaction | 112
  Any Injection site Erythema (N = 129) | 61
  Grade 3 Erythema (≥5 cm; N = 129) | 4
  Any Injection site Swelling (N = 129) | 40
  Grade 3 Swelling (≥5 cm; N = 129) | 2
  Any injection site Pain (N = 129) | 102
  Grade 3 Pain (Incapacitating; N = 129) | 1
  Any extensive swelling of vaccinated limb (N=129) | 0
  Grade 3 extensive swelling of vaccinated limb N129 | 0
  Any Solicited Systemic Reaction (N = 130) | 63
  Any Fever (N = 130) | 14
  Grade 3 Fever (> 39.0°C; N = 130) | 2
  Any Headache (N = 130) | 28
  Grade 3 Headache (Prevents daily activities; N=130 | 1
  Any Myalgia (N = 130) | 46
  Grade 3 Myalgia (Prevents daily activities; N=130) | 0
  Any Malaise (N = 130) | 27
  Grade 3 Malaise (Prevents daily activities; N=130) | 0

ADVERSE EVENTS:
Time Frame: Adverse events data were collected from following vaccination (Day 0) for up to 1 month post-vaccination.
Arm/Group | ADACEL POLIO Vaccine Study Group
Serious Adverse Events (participants affected / at risk) | 2/132
Other Adverse Events (participants affected / at risk) | 102/132
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ADACEL POLIO Vaccine Study Group (N=132)
Gastroenteritis (Infections and infestations) | 1 (1)
Thermal burn (Injury, poisoning and procedural complications) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ADACEL POLIO Vaccine Study Group (N=132)
Injection Site Pain (General disorders) | 102 (102)
Injection site Erythema (General disorders) | 61 (61)
Fever (General disorders) | 14 (14)
Malaise (General disorders) | 27 (27)
Injection Site Swelling (General disorders) | 40 (40)
Myalgia (Musculoskeletal and connective tissue disorders) | 46 (46)
Headache (Nervous system disorders) | 28 (28)
Nasopharyngitis (Infections and infestations) | 19 (19)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor must have the opportunity to review at least 60 days prior to submission for publication or presentation. If review indicates that potentially patentable subject matter would be disclosed, publication or public disclosure may be delayed for a maximum of an additional 60 days to allow for filing the necessary patent applications